CLINICAL TRIAL: NCT03759574
Title: Pathophysiologic Hemodynamics After Primary Unilateral Total Hip Arthroplasty
Brief Title: Pathophysiologic Hemodynamics After Primary Unilateral Total Hip Arthroplasty (THA)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Kehlet, Henrik, M.D., Ph.D. (Individual)
Responsible Party: Principal Investigator, Ana-Marija Hristovska, Prinicial Investigator, Medical Doctor, PhD-student, Hvidovre University Hospital
Other Study IDs: H-18052195
Record Dates: First submitted 2018-11-28; First posted 2018-11-30 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Orthostatic Intolerance; Orthostatic Hypotension; Postoperative Complications
Keywords: Orthostatic Intolerance; Orthostatic Hypotension
MeSH Terms: conditions — Orthostatic Intolerance; Hypotension, Orthostatic; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Orthostatic intolerant (OI): Patients that experience symptoms of orthostatic intolerance (dizziness, nausea, vomiting, blurry vision or syncope) or orthostatic hypotension (fall in systolic pressure > 20 mmHg and/or diastolic pressure > 10 mmHg) during mobilisation
- Orthostatic tolerant (OT): Patients that do not experience symptoms of orthostatic intolerance (dizziness, nausea, vomiting, blurry vision or syncope) or orthostatic hypotension (fall in systolic pressure > 20 mmHg and/or diastolic pressure > 10 mmHg) during mobilisation

SUMMARY:
Incidence and pathophysiologic hemodynamics of orthostatic intolerance and orthostatic hypotension in patients undergoing unilateral THA

DETAILED DESCRIPTION:
Early postoperative mobilization is a cornerstone in the so-called fast track multimodal perioperative approach and is essential in preventing postoperative morbidity and reducing hospital length-of-stay. Intact orthostatic blood pressure regulation is essential for early postoperative mobilization. However, early postoperative mobilization can be delayed due to postoperative orthostatic hypotension (POH) defined as a fall in systolic pressure > 20 mmHg and/or diastolic pressure > 10 mmHg or due to postoperative orthostatic intolerance (POI), characterized by dizziness, nausea, vomiting, blurred vision or syncope during mobilization. Although these conditions are well-known clinical problems that can delay early mobilization, relatively few data are available on pathophysiological mechanisms and possible treatments.

Several prospective studies with standardized mobilization procedures have already established that the incidence of POI and POH after THA is 38-42% at 6 hours after surgery.

Previous studies on patients undergoing prostatectomy and THA have also demonstrated that attenuated vasopressor response and a concomitant reduction in cardiac output (CO) and cerebral perfusion during postural changes after surgery contributes to POI and POH. Strategies aiming to reduce the incidence of POI and POH by pain management, vasoconstrictive treatment with alpha-1 receptor agonist, optimized fluid management with goal-directed fluid therapy and reduction of surgical stress-response with pre-operative high-dose glucocorticoid did not solve the problem.

The precise pathophysiological mechanisms of POI and POH remain to be elucidated and this is therefore the aim of the current prospective observational study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Written informed consent
* Patients that speak and understand Danish
* Patients undergoing primary unilateral total hip arthroplasty in spinal anesthesia in standardized fast-track setting

Exclusion Criteria:

* Alcohol and drug abuse
* Cognitive dysfunction
* History of orthostatic hypotension
* Use of anxiolytic or antipsychotic drugs
* Use of opioids
* Use of following vasodilator antihypertensive drugs: beta-blockers, angiotensin converting enzyme inhibitors (ACEI), angiotensin 2 receptor blockers (ARBs), calcium channel blockers
* Use of loop diuretics, thiazid diuretics and potassium-sparing diuretics
* Use of Gabapentin
* Arrhythmias or heart failure
* Diabetes mellitus type I
* Diabetes mellitus type II
* History of following diseases in the autonomic nervous system: Parkinson disease, multiple sclerosis, autonomic neuropathies
* History of cerebral apoplexy or transitory cerebral ischemia
* Dementia
* American Society of Anesthesiologists (ASA) score ≥ 4

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing primary unilateral total hip arthroplasty in spinal anesthesia in standardized fast-track setting
Sampling Method: Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2019-03-18 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-05-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of orthostatic intolerance | 6 hours postoperatively
  Symptoms of orthostatic intolerance: dizziness, nausea, vomiting, blurry vision or syncope during mobilization
Incidence of orthostatic hypotension | 6 hours postoperatively
  Orthostatic hypotension is defined as a fall in systolic pressure > 20 mmHg and/or diastolic pressure > 10 mmHg during mobilization

SECONDARY OUTCOMES:
Changes in systolic arterial pressure (SAP) during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured in mmHg
Changes in diastolic arterial pressure (DAP) during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured in mmHg
Changes in mean arterial pressure (MAP) during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured in mmHg
Changes in systemic vascular resistance (SVR) during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured in mmHg⋅min⋅mL-1
Changes in cardiac output (CO) during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured in mL/min
Changes in stroke volume (SV) during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured in mL
Changes in heart rate variability (HRV) during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured in ms
Changes in baroreflex sensitivity (BRS) during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured in ms/mmHg
Changes in peripheral perfusion index (PPI) during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured in arbitrary units (AU)
Changes in cerebral perfusion (ScO2) during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured in %
Changes in muscular perfusion (SmO2) during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured in %
Changes in total blood volume (TBV) | Preoperatively, 6 and 24 hours postoperatively
  Measured in mL
Changes in erythrocyte volume (ECV) | Preoperatively, 6 and 24 hours postoperatively
  Measured in mL
Changes in plasma volume (PV) | Preoperatively, 6 and 24 hours postoperatively
  Measured in mL
Changes in hematocrit | Preoperatively, 6 and 24 hours postoperatively
  Measured in %
Changes in haemoglobin (Hgb) concentration | Preoperatively, 6 and 24 hours postoperatively
  Measured in millimoles/L
Changes in C-Reactive Protein | Preoperatively, 6 and 24 hours postoperatively
  Measured in mg/L

OTHER OUTCOMES:
Pain score | Preoperatively, 6 and 24 hours postoperatively
  Measured by verbal rating scale (VRS) from 0 to 10 (0 = no pain, 10 = worse pain imaginable)
Estimated bleeding | Intraoperatively, 6 and 24 hours postoperatively
  Measured in mL
Opioid use | 6 and 24 hours postoperatively
  Measured in mg
Cumulative fluid administration and losses | Intraoperatively, 6 and 24 hours postoperatively
  Measured in mg

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jans O, Bundgaard-Nielsen M, Solgaard S, Johansson PI, Kehlet H. Orthostatic intolerance during early mobilization after fast-track hip arthroplasty. Br J Anaesth. 2012 Mar;108(3):436-43. doi: 10.1093/bja/aer403. Epub 2011 Dec 15. PMID 22174345
- [Background] Lindberg-Larsen V, Petersen PB, Jans O, Beck T, Kehlet H. Effect of pre-operative methylprednisolone on orthostatic hypotension during early mobilization after total hip arthroplasty. Acta Anaesthesiol Scand. 2018 Aug;62(7):882-892. doi: 10.1111/aas.13108. Epub 2018 Mar 24. PMID 29573263
- [Background] Jans O, Mehlsen J, Kjaersgaard-Andersen P, Husted H, Solgaard S, Josiassen J, Lunn TH, Kehlet H. Oral Midodrine Hydrochloride for Prevention of Orthostatic Hypotension during Early Mobilization after Hip Arthroplasty: A Randomized, Double-blind, Placebo-controlled Trial. Anesthesiology. 2015 Dec;123(6):1292-300. doi: 10.1097/ALN.0000000000000890. PMID 26492477
- [Background] Bundgaard-Nielsen M, Jans O, Muller RG, Korshin A, Ruhnau B, Bie P, Secher NH, Kehlet H. Does goal-directed fluid therapy affect postoperative orthostatic intolerance?: A randomized trial. Anesthesiology. 2013 Oct;119(4):813-23. doi: 10.1097/ALN.0b013e31829ce4ea. PMID 23756453
- [Background] Jans O, Kehlet H. Postoperative orthostatic intolerance: a common perioperative problem with few available solutions. Can J Anaesth. 2017 Jan;64(1):10-15. doi: 10.1007/s12630-016-0734-7. Epub 2016 Sep 14. No abstract available. PMID 27638295